CLINICAL TRIAL: NCT07051265
Title: Effect of Transcutaneous Electrical Nerve Stimulation (TENS) or Acupressure on Pain in Patients With Head and Neck Cancer
Brief Title: Effect of Transcutaneous Electrical Nerve Stimulation or Acupressure on Pain in Patients With Head and Neck Cancer
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Li-Ying Lin, Nursing Department Supervisor, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KSVGH25-CT4-03
Record Dates: First submitted 2025-05-25; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Head and Neck Cancer; Cancer Pain
Keywords: Transcutaneous Electrical Nerve Stimulation; Acupressure; Cancer pain; Head and neck cancer; Quality of life; emotional distress
MeSH Terms: conditions — Head and Neck Neoplasms; Cancer Pain | interventions — Transcutaneous Electric Nerve Stimulation; Acupressure

STUDY DESIGN:
Intervention Model Description: The patients with head and neck cancer were randomly assigned to an intervention group or a control group using computer random numbers. The intervention group was further divided into two groups: transcutaneous electrical nerve stimulation intervention and acupoint pressing measures.
  The transcutaneous electrical stimulation group used a transcutaneous electrical nerve stimulator daily, with electrode patches attached to the unilateral Hegu and Lieque points for 20 minutes of 80-100 Hz TAES stimulation, three times a day, and the electrical stimulation was adjusted to a level that the subjects felt was comfortable. The acupressure group also selected Hegu and Lieque points for the treatment, placed the acupoint stickers on the acupoints of both hands, and pressed each acupoint with the thumb and index finger for 1 minute, 3 times a day, each time for about 4 minutes.
  The control group took the original analgesics and did not receive any acupoint stimulation.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): Maintain normal treatment without any intervention
- Transcutaneous Electrical Nerve Stimulation (TENS) (Experimental): The transcutaneous electrical stimulation group used a transcutaneous electrical nerve stimulator daily, with electrode patches attached to the unilateral Hegu and Lieque points respectively, providing 20 minutes of 80-100 HZ TENS, 3 times a day, and the electrical stimulation was adjusted to a level that the subjects felt was comfortable.
  Interventions: Behavioral: Transcutaneous Electrical Nerve Stimulation (TENS)
- Acupressure (Experimental): The acupressure group selected Hegu and Lieque points for the treatment, placed the acupoint stickers on the acupoints of both hands, and pressed each acupoint with the thumb and index finger for 1 minute, 3 times a day, each time for about 4 minutes.
  Interventions: Behavioral: Acupressure

INTERVENTIONS:
Behavioral: Transcutaneous Electrical Nerve Stimulation (TENS) — Participants received TENS therapy at two specific acupoints - Hegu (LI4) and Lieque (LU7). Surface electrodes were placed over the acupoints, and stimulation was delivered using a standard TENS device.
  Arms: Transcutaneous Electrical Nerve Stimulation (TENS)
Behavioral: Acupressure — The acupressure group placed the acupoint patches on the Hegu and Lieque points on both hands and pressed each acupoint with the index finger and thumb for 1 minute, 3 times a day, each time for about 4 minutes.
  Arms: Acupressure

SUMMARY:
This clinical trial aims to evaluate the effectiveness of transcutaneous electrical nerve stimulation (TENS), acupressure intervention, or standard care (control group) for pain management in participants hospitalized with head and neck cancer. This study aims to answer the following questions:

* Is TENS or acupressure intervention effective in reducing pain in participants hospitalized with head and neck cancer compared with the control group?
* Does TENS or acupressure intervention improve psychological distress (measured by the Brief Health Inventory (BMI)) in these participants?
* Does TENS or acupressure intervention improve the quality of life of participants hospitalized with head and neck cancer? Researchers will compare the effects of TENS, acupressure, and standard care to assess the effects of each group on pain, psychological distress (measured by the Brief Health Inventory (BMI)), and quality of life.

DETAILED DESCRIPTION:
Study Procedure:

A. If the participant agrees to participate in the study and signs the informed consent form, the researcher will ask them to complete a questionnaire. The questionnaire includes basic demographic information, pain level, emotional distress (Brief Symptom Rating Scale), and quality of life survey. It takes about 10 minutes to complete the questionnaire.

B. Participants will be randomly assigned to one of the following three groups:

* Transcutaneous electrical nerve stimulation (TENS) combined with standard treatment
* Acupressure combined with standard treatment
* Standard treatment (control group) C. Before and after daily intervention, all three groups of participants will complete a numerical rating scale (0-10 points) to assess pain intensity, and their vital signs will be recorded.

D. After one week of intervention, every week thereafter, and before discharge, participants will complete a numerical rating scale (0-10 points), the Brief Symptom Rating Scale (BSRS), and the World Health Organization Quality of Life Brief Form (WHOQOL-BREF).

Possible side effects and how to cope with them:

• TENS or acupressure: Participants may experience soreness, tingling, pressure, or mild pain when using TENS or acupressure to treat the Hegu (LI4) and Lieque (LU7) points. These are normal reactions and are generally well tolerated. No studies have shown any harmful side effects from stimulating these points. If discomfort is too great, the intensity of stimulation can be adjusted.

• Risks to participants: Participants can stop at any time if they feel discomfort during the study. Participants can also contact the study's emergency contact for assistance.

Expected benefits:

Previous research and traditional practices have shown that acupressure on the Hegu (LI4) and Lieque (LU7) points may help regulate the flow of Qi and blood, enhance lung function, improve blood circulation, and relieve pain and discomfort. While researchers cannot guarantee that this study will benefit participants, acupressure may help healthcare professionals better understand how to support clinical inpatients (non-participants) and may benefit others in the future.

Participant privacy is protected: Researchers will only collect information necessary for this study. All participant personal information and questionnaire responses will remain confidential. Participants' names and personal identifying information will not be used; instead, researchers will assign participants a code to ensure that the participant's identity remains anonymous in all records.

ELIGIBILITY:
Participant inclusion criteria:

1. Age ≥ 20 years old
2. Inpatients diagnosed with head and neck cancer
3. Conscious and able to communicate in Mandarin and Taiwanese
4. Suffering from pain problems and requiring pain medication
5. Participants agree to participate in this study.

Participant exclusion criteria:

1. Those with nerve conduction disorders
2. Pregnant women
3. Those whose pain is not caused by tumors
4. Those with a history of epilepsy
5. Those with skin infections
6. Those who are allergic to the patch
7. Those with implanted devices such as pacemakers
8. Those who still disagree with the study content and are unable to cooperate with the researchers after the researchers' explanation.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale | Daily for up to 14 days
  A self-reporting tool to assess subjective experience (such as symptoms, feelings and attitudes). On a 10 mm straight line (0-10 points from left to right), the far left side represents no pain (0 points) and the far right side represents extreme pain (10 points). The higher the pain score, the more severe the pain. The subjects were asked to describe the pain intensity themselves. This method has a good intraclass correlation coefficient for pain assessment (ICC=0.99). After the subjects started the trial, they were required to fill in the numerical scale three times a day (9 am, 12 pm and 4 pm). Each filling was divided into before the intervention (pretest) and after the intervention (posttest). Therefore, the pain index will be recorded 6 times a day. The numerical scale will be filled in until they are discharged from the hospital or transferred to another ward (whichever comes first).

SECONDARY OUTCOMES:
Brief Symptom Rating Scale | Baseline, Day 7, and Day 14 or until discharge/transfer, whichever occurred first.
  The Brief Symptom Rating Scale (BSRS-5) compiled by Professor Li Mingbin can quickly understand an individual's psychological care needs. The BSRS consists of 5 questions (measuring anxiety, anger, depression, low self-esteem and insomnia) and 1 additional question. Participants used a 5-point Likert scale (0-4 points), where 0 represented "not at all", 1 represented "mild", 2 represented "moderate", 3 represented "severe", and 4 represented "very severe", with a total score of 0-20 points. The higher the score, the more severe the psychological distress. The Cronbach's α value measured for the sample in this study was 0.829, which has a high internal consistency reliability. Participants will complete the BSRS-5 assessment once at the beginning of the program, and then complete the follow-up once a week (start day (pre-test) + 7 days, 14 days, 28 days, etc.) until they are discharged from the hospital or transferred to another ward (whichever comes first).
The Taiwanese version of the World Health Organization Quality of Life Questionnaire | Baseline, Day 7, and Day 14 or until discharge/transfer, whichever occurred first.
  The World Health Organization Quality of Life Questionnaire (WHOQOL BREF) developed by Yao Qizhi was used to measure the overall quality of life, general health status and 24 aspects of quality of life, which are divided into four categories: "physical health (covering the original physical and independence categories), psychological (covering the original psychological and spiritual/religious/personal belief categories), social relationships and environment". The scale consists of 28 questions, each with a score range of 1-5 points, and a total score of 28-140 points. The higher the score, the better the quality of life. Participants will complete the World Health Organization Quality of Life Questionnaire Taiwan Version (pre-test) once after the start of the program, and then complete it once a week (starting day + 7 days, 14 days, 28 days, etc.) until they were discharged or transferred to other wards whichever came first.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Ling Li, Principal Investigator — Supervision
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bijur PE, Silver W, Gallagher EJ. Reliability of the visual analog scale for measurement of acute pain. Acad Emerg Med. 2001 Dec;8(12):1153-7. doi: 10.1111/j.1553-2712.2001.tb01132.x. PMID 11733293
- [Background] Brant JM, Eaton LH, Irwin MM. Cancer-Related Pain: Assessment and Management With Putting Evidence Into Practice Interventions . Clin J Oncol Nurs. 2017 Jun 1;21(3 Suppl):4-7. doi: 10.1188/17.CJON.S3.4-7. PMID 28524908
- [Background] Chou YH, Yeh ML, Huang TS, Hsu H. Acupoint stimulation improves pain and quality of life in head and neck cancer patients with chemoradiotherapy: A randomized controlled trial. Asia Pac J Oncol Nurs. 2021 Dec 25;9(1):61-68. doi: 10.1016/j.apjon.2021.11.002. eCollection 2022 Jan. PMID 35528798
- [Background] Ge L, Wang Q, He Y, Wu D, Zhou Q, Xu N, Yang K, Chen Y, Zhang AL, Hua H, Huang J, Hui KK, Liang F, Wang L, Xu B, Yang Y, Zhang W, Zhao B, Zhu B, Guo X, Xue CC, Zhang H; International Trustworthy traditional Chinese Medicine Recommendations (TCM Recs) Working Group. Acupuncture for cancer pain: an evidence-based clinical practice guideline. Chin Med. 2022 Jan 5;17(1):8. doi: 10.1186/s13020-021-00558-4. PMID 34983587
- [Background] Gift AG. Visual analogue scales: measurement of subjective phenomena. Nurs Res. 1989 Sep-Oct;38(5):286-8. No abstract available. PMID 2678015
- [Background] Harrington CB, Hansen JA, Moskowitz M, Todd BL, Feuerstein M. It's not over when it's over: long-term symptoms in cancer survivors--a systematic review. Int J Psychiatry Med. 2010;40(2):163-81. doi: 10.2190/PM.40.2.c. PMID 20848873
- [Background] Hermann GM, Iovoli AJ, Platek AJ, Wang C, Miller A, Attwood K, Bourgeois DJ, Singh AK. A single-institution, randomized, pilot study evaluating the efficacy of gabapentin and methadone for patients undergoing chemoradiation for head and neck squamous cell cancer. Cancer. 2020 Apr 1;126(7):1480-1491. doi: 10.1002/cncr.32676. Epub 2019 Dec 23. PMID 31869451
- [Background] He Y, Guo X, May BH, Zhang AL, Liu Y, Lu C, Mao JJ, Xue CC, Zhang H. Clinical Evidence for Association of Acupuncture and Acupressure With Improved Cancer Pain: A Systematic Review and Meta-Analysis. JAMA Oncol. 2020 Feb 1;6(2):271-278. doi: 10.1001/jamaoncol.2019.5233. PMID 31855257
- [Background] Kasasbeh MAM, McCabe C, Payne S. Cancer-related pain management: A review of knowledge and attitudes of healthcare professionals. Eur J Cancer Care (Engl). 2017 Nov;26(6). doi: 10.1111/ecc.12625. Epub 2016 Dec 27. PMID 28026070
- [Background] Kramer S, Newcomb M, Hessler J, Siddiqui F. Prophylactic versus reactive PEG tube placement in head and neck cancer. Otolaryngol Head Neck Surg. 2014 Mar;150(3):407-12. doi: 10.1177/0194599813517081. Epub 2013 Dec 31. PMID 24381015
- [Background] Lee JE, Anderson CM, Perkhounkova Y, Sleeuwenhoek BM, Louison RR. Transcutaneous Electrical Nerve Stimulation Reduces Resting Pain in Head and Neck Cancer Patients: A Randomized and Placebo-Controlled Double-Blind Pilot Study. Cancer Nurs. 2019 May/Jun;42(3):218-228. doi: 10.1097/NCC.0000000000000594. PMID 29649082
- [Background] Lee MB, Lee YJ, Yen LL, Lin MH, Lue BH. Reliability and validity of using a Brief Psychiatric Symptom Rating Scale in clinical practice. J Formos Med Assoc. 1990 Dec;89(12):1081-7. PMID 1982678
- [Background] Lee MB, Liao SC, Lee YJ, Wu CH, Tseng MC, Gau SF, Rau CL. Development and verification of validity and reliability of a short screening instrument to identify psychiatric morbidity. J Formos Med Assoc. 2003 Oct;102(10):687-94. PMID 14691593
- [Background] Loh J, Gulati A. The use of transcutaneous electrical nerve stimulation (TENS) in a major cancer center for the treatment of severe cancer-related pain and associated disability. Pain Med. 2015 Jun;16(6):1204-10. doi: 10.1111/pme.12038. Epub 2013 Feb 25. PMID 23438255
- [Background] Maindet C, Burnod A, Minello C, George B, Allano G, Lemaire A. Strategies of complementary and integrative therapies in cancer-related pain-attaining exhaustive cancer pain management. Support Care Cancer. 2019 Aug;27(8):3119-3132. doi: 10.1007/s00520-019-04829-7. Epub 2019 May 11. PMID 31076901
- [Background] Melzack R, Wall PD. Pain mechanisms: a new theory. Science. 1965 Nov 19;150(3699):971-9. doi: 10.1126/science.150.3699.971. No abstract available. PMID 5320816
- [Background] Sluka KA, Vance CG, Lisi TL. High-frequency, but not low-frequency, transcutaneous electrical nerve stimulation reduces aspartate and glutamate release in the spinal cord dorsal horn. J Neurochem. 2005 Dec;95(6):1794-801. doi: 10.1111/j.1471-4159.2005.03511.x. Epub 2005 Oct 17. PMID 16236028
- [Background] Strom T, Trotti AM, Kish J, Rao NG, McCaffrey J, Padhya TA, Lin HY, Fulp W, Caudell JJ. Risk factors for percutaneous endoscopic gastrostomy tube placement during chemoradiotherapy for oropharyngeal cancer. JAMA Otolaryngol Head Neck Surg. 2013 Nov;139(11):1242-6. doi: 10.1001/jamaoto.2013.5193. PMID 24136493
- [Background] Wong PC, Dodd MJ, Miaskowski C, Paul SM, Bank KA, Shiba GH, Facione N. Mucositis pain induced by radiation therapy: prevalence, severity, and use of self-care behaviors. J Pain Symptom Manage. 2006 Jul;32(1):27-37. doi: 10.1016/j.jpainsymman.2005.12.020. PMID 16824982
- [Background] Yao G, Chung CW, Yu CF, Wang JD. Development and verification of validity and reliability of the WHOQOL-BREF Taiwan version. J Formos Med Assoc. 2002 May;101(5):342-51. PMID 12101852
- [Background] Shen WC, Chen JS, Shao YY, Lee KD, Chiou TJ, Sung YC, Rau KM, Yen CJ, Liao YM, Liu TC, Wu MF, Lee MY, Yu MS, Hwang WL, Lai PY, Chang CS, Chou WC, Hsieh RK. Impact of Undertreatment of Cancer Pain With Analgesic Drugs on Patient Outcomes: A Nationwide Survey of Outpatient Cancer Patient Care in Taiwan. J Pain Symptom Manage. 2017 Jul;54(1):55-65.e1. doi: 10.1016/j.jpainsymman.2017.02.018. Epub 2017 May 4. PMID 28479410
- See also: Development and Applications of the WHOQOL-Taiwan Version — https://doi.org/10.6320/FJM.2002.6(2).09
- See also: Pain mechanisms: A new theory: A gate control system modulates sensory input from the skin before it evokes pain perception and response — https://doi.org/10.1016/S1082-3174(96)80062-6
- See also: Cancer Facts & Figures 2018 — https://www.cancer.org/research/cancer-facts-statistics/all-cancer-facts-figures/cancer-facts-figures-2018.html
- See also: Transcutaneous Electrical Nerve Stimulation in Patients with CancerRelated Pain: A Systematic Review — https://saudijournals.com/media/articles/SJBR-47-270-278.pdf
- See also: The Experiences and Outcomes of Promoting Cancer Painless College at a Medical Center — https://doi.org/10.6880/TJON.201903/SP_19.15
- See also: Effects of an Acupoint Intervention on Improving Fatigue and Heart Rate Variability in Head and Neck Cancer Patients Receiving Concurrent Chemoradiotherapy — https://doi.org/10.6224/JN.201906_66(3).07
- See also: A review on the psychometric properties of the WHOQOL-BREF — https://doi.org/10.6288/TJPH.201912_38(6).108087
- See also: The incidence of the top ten cancers — https://www.gender.ey.gov.tw/gecdb/Stat_Statistics_DetailData.aspx?sn=nLF9GdMD%2B%2Bv41SsobdVgKw%3D%3D